CLINICAL TRIAL: NCT02269852
Title: A Single-centered, Open-labeled, Phase 4 Study of a Northern Hemisphere 2013-2014 Seasonal Trivalent Influenza Inactivated Vaccine, Anflu®
Brief Title: The Immunogenicity and Safety of 2013-2014 Seasonal Trivalent Influenza Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO-INF-4013
Record Dates: First submitted 2014-10-08; First posted 2014-10-21 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Influenza
Keywords: seasonal trivalent inactivated influenza vaccine; immunogenicity; safety; cross-reactivity; Northern hemisphere 2013-2014 formulation
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- trivalent seasonal influenza vaccine (Experimental): Northern hemisphere 2013-2014 trivalent seasonal influenza vaccine
  * 60 infants: two-dose regimen with a 28-day interval;
  * 60 adults: single-dose regimen;
  * 60 seniors: single-dose regimen;
  Interventions: Biological: trivalent seasonal influenza vaccine

INTERVENTIONS:
Biological: trivalent seasonal influenza vaccine — * Infants: 0.25 ml/ dose;
  * Adults: 0.5 ml/ dose;
  * Seniors: 0.5 ml/ dose;
  Other Names: Anflu®

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of Northern hemisphere 2013-2014 seasonal trivalent inactivated influenza vaccine in 60 healthy infants aged 6-35 months old, 60 healthy adults aged 18-60 years old, and 60 healthy seniors aged > 60 years.

ELIGIBILITY:
For adults and seniors:

Inclusion Criteria:

* Healthy adults aged 18-60 years old, and healthy seniors aged > 60 years old;
* Without vaccination history of seasonal split influenza vaccine in the recent 3 years
* No traveling plan during the study period of this trial;
* Be able to understand and sign the informed consent;

Exclusion Criteria:

* Allergic to egg products or any ingredient of the study vaccine;
* Fever, influenza or acute illness on the vaccination day;
* Acute stage of chronic illness;
* Malignant tumor;
* Immunodeficiency, includes HIV infection;
* Guillain-Barre syndrome;
* Administration of live attenuated vaccine within the previous 14 days;
* Administration of subunit or inactivated vaccine within the previous 7 days;
* Planned to participate in any other clinical trial of drug or vaccine during this study;
* Received immunesuppressive treatment within the previous month, or planned for such treatment during this study;
* Pregnant, or planning pregnancy;
* Axillary temperature > 37.0℃;
* Any other factors that, in the judgment of the investigator, is unsuitable for this study;

For infants:

Inclusion Criteria:

* Healthy male or female aged between 6 and 35 months;
* Full-term birth, birth weight 2,500 grams or more;
* Provided birth certification or vaccination card
* Parent or legal guardian is able to understand and sign the informed consent;

Exclusion Criteria:

* Received seasonal influenza vaccine after June 30, 2012;
* Acute infection within the previous week;
* Allergy history, or allergic to any ingredient of the study vaccine, such as egg;
* History of serious adverse reaction (SAR) to vaccine;
* Autoimmune disease or immune deficiency, or administration of immunosuppressive therapy, cell toxic therapy, or inhaled corticosteroid within the previous 6 months;
* Congenital malformations, developmental disorder or serious chronic disease;
* Unstable condition of asthma and administration of corticosteroid in the most recent two years;
* Coagulation abnormalities or disorders;
* History/ family history of infantile convulsion, epilepsy, cerebropathy, or mental disease;
* Without spleen;
* Severe neurological diseases, such as Guillain-Barre syndrome;
* Administration of blood products or investigational drug within the previous month;
* Administration of live attenuated vaccine within the previous 14 days;
* Administration of subunit or inactivated vaccine within the previous 7 days;
* Received treatment for allergy within the previous 14 days;
* on-going anti-tuberculosis therapy;
* Axillary temperature > 37.0℃ immediately before vaccination;
* any other factors that, in the judgment of the investigator, is unsuitable for this study;

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The immunogenicity of 2013-2014 seasonal trivalent vaccine (TIV) in adults and seniors | 21 days after vaccination
  To evaluate the immune responses to each antigen of the 2013-2014 seasonal TIV in adults and seniors by detection of hemagglutination inhibition (HI) antibody titer

SECONDARY OUTCOMES:
The incidences of adverse events (AEs) in infants, adults and seniors | Day 0 - day 35
  After each injection, a 30-minute safety observation was conducted immediately, and the body temperature, occurrence of solicited local and general AEs within 72 hours were collected. Unsolicited AEs of adults and seniors were collected until day 21, and those of infants were collected until day 35. Each AE case was reviewed by the investigator to determine whether or not it was an adverse reaction (related to the vaccination).
The cross-reactivity of 2013-2014 seasonal TIV in adults and seniors against influenza B Victoria lineage virus and the avian influenza A(H7N9) virus | 21 days after vaccination
  To evaluate the cross-reactivity of 2013-2014 seasonal TIV in adults and seniors against influenza B Victoria lineage virus (not in the vaccine formulation) and the avian influenza A(H7N9) virus by detection of HI antibody titer

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Gang Shen, Principal Investigator — Anhui Center for Diseases Control and Prevention
Locations (1):
- Guzhen Center for Diseases Control and Prevention, Bengbu, Anhui, China

REFERENCES:
- [Derived] Shen Y, Hu Y, Meng F, Du W, Li W, Song Y, Ji X, Huo L, Fu Z, Yin W. Safety, immunogenicity and cross-reactivity of a Northern hemisphere 2013-2014 seasonal trivalent inactivated split influenza virus vaccine, Anflu(R). Hum Vaccin Immunother. 2016 May 3;12(5):1229-34. doi: 10.1080/21645515.2015.1123357. Epub 2016 Mar 2. PMID 26934750